CLINICAL TRIAL: NCT02070211
Title: Indicated Prevention With Long-chain Polyunsaturated Omega-3 Fatty Acids in Patients With 22q11 Microdeletion Syndrome Genetically at High Risk for Psychosis: A Randomised, Double Blind, Placebo-controlled Treatment Trial.
Brief Title: Indicated Prevention With Long-chain Polyunsaturated Omega-3 Fatty Acids in Patients With 22q11 Microdeletion Syndrome.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); Orygen (Other)
Responsible Party: Principal Investigator, Marco Armando, MD, PhD, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: APS 1; 21278 (Other Grant/Funding Number: NARSAD Young Investigator Grant)
Record Dates: First submitted 2014-02-17; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: 22q11 Deletion Syndrome
Keywords: Psychotic Disorder; 22q11 Deletion Syndrome; Fatty Acids, Omega-3
MeSH Terms: conditions — 22q11 Deletion Syndrome; Psychotic Disorders | interventions — Fish Oils; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- omega-3 PUFAs in add on to standard care (Experimental): omega-3 PUFA supplementation as an adjunct to non-neuroleptic, standard therapy in individuals with 22q11DS and UHR criteria for psychosis
  Interventions: Dietary Supplement: omega-3 PUFAs; Other: Standard care
- Placebo in add on to standard care (Placebo Comparator): Placebo made by paraffin oil (not absorbed by the gastrointestinal tract) as an adjunct to non-neuroleptic, standard therapy in individuals with 22q11DS and UHR criteria for psychosis
  Interventions: Other: Standard care; Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: omega-3 PUFAs — 4 capsules (2 in the morning; 2 in the evening) for a period of 12 weeks. The active treatment is a supplement of yellow gelatine 0.625 g capsules containing concentrated marine fish oil. The daily dose of 4 capsules will provide approximately 700 mg of eicosapentaenoic acid (EPA, 20:5n3), 480 mg of docosahexaenoic acid (DHA, 22:6n3), and 7.6 mg of Vitamin E.
  Other Names: fish oil; poly unsaturated fatty acids
  Arms: omega-3 PUFAs in add on to standard care
Other: Standard care — Standard care includes management by a psychiatrist or resident psychiatrist and non-neuroleptic pharmacotherapy as clinically indicated. Specifically, Cognitive-behavioural therapy (CBT) embedded within case management will be administered. The CBT will be based on the models developed at the PACE Clinic in Melbourne, in the EDIE trial, and in Cologne, as these have proven to be effective in RCTs. The number of sessions delivered will be captured for each client. In addition, fidelity will be monitored by therapists rating their own sessions on an established checklist of therapeutic interventions.
Dietary Supplement: placebo — 4 capsules of 0.7g of paraffin oil (which is not absorbed by the gastrointestinal tract) per day.
  Arms: Placebo in add on to standard care

SUMMARY:
The purpose of the present trial is to investigate the effects of omega-3 PUFAs in individuals aged 12-26 years with 22q11DS at ultra-high risk for developing a first episode of psychosis.

DETAILED DESCRIPTION:
We will use a prospective, randomized, double-blind, placebo-controlled, single-centre study design. Eighty individuals aged 12-26 will be randomly assigned in two treatment conditions (40 in each arm) at the Department of Neuroscience, Children Hospital Bambino Gesù, Rome, Italy. Randomisation will be arranged by the Clinical Trials Department of the same hospital. Participants will receive 4 capsules (2 in the morning; 2 in the evening) for a period of 12 weeks. The active treatment is a supplement of yellow gelatine 0.625 g capsules containing concentrated marine fish oil. The daily dose of 4 capsules will provide approximately 700 mg of eicosapentaenoic acid (EPA, 20:5n3), 480 mg of docosahexaenoic acid (DHA, 22:6n3), and 7.6 mg of Vitamin E. Vitamin E is added as an antioxidant to fish oil capsules to stabilize highly unsaturated fatty acids. Participants will receive either 4 capsules of 0.7g marine fish oil or 4 capsules of 0.7g of paraffin oil (which is not absorbed by the gastrointestinal tract) per day. The daily dose of omega-3 PUFAs is based on our previous trail (Amminger et al., 2010).

All patients will receive standard treatment, which includes management by a psychiatrist or resident psychiatrist and non-neuroleptic pharmacotherapy as clinically indicated. Specifically, Cognitive-behavioural therapy (CBT) embedded within case management will be administered. The CBT will be based on the models developed at the PACE Clinic in Melbourne, in the EDIE trial, and in Cologne, as these have proven to be effective in RCTs. The number of sessions delivered will be captured for each client. In addition, fidelity will be monitored by therapists rating their own sessions on an established checklist of therapeutic interventions. Any additional psychosocial interventions delivered will also be documented. The case management component will consist of therapists addressing current interpersonal and social issues and providing practical help. 6 - 20 CBCM sessions will be provided within the first 6 months.

Hypotheses:

1. Omega-3 PUFAs have a positive effect on clinical course and outcome in UHR+22q11DS individuals

   Specifically that at 12 months follow-up:
   * The transition to psychosis rate is significantly lower in the omega-3 PUFA group
   * Ratings on CAARMS, PANSS, MADRS, GAF improve significantly more in the omega-3 PUFA group
   * Neuropsychological functioning is significantly better in the omega-3 PUFA group.
2. Lipid metabolism characteristics described in schizophrenia will be more prevalent in individuals who make transition to psychosis

   * Reduced omega-3 PUFAs and reduced nervonic acid (Amminger et al., 2011) and increased PLA2 activity at baseline characterize individuals who develop psychosis
   * PLA2 activity will significantly decrease pre/post treatment in the omega-3 PUFA group

ELIGIBILITY:
Inclusion Criteria:

* written informed consent (for individuals under 18 written informed consent of parents is required);
* age between 12 and 26 years;
* UHR as classified by the CAARMS (Yung et al., 2005);
* genetic diagnosis of 22q11DS

Exclusion Criteria:

* acute suicidal behaviour (score of 6 on CAARMS item 7.3) or aggressive behaviour (score of 6 on CAARMS item 5.4);
* Drug abuse that contributed decisively to the presentation of the index episode, (dependency on morphine, cocaine, amphetamine, but not THC);
* Alcohol abuse if considered as major problem;
* Epilepsy; 5./IQ<70);
* Pregnancy and lactation;
* Previous history of antipsychotic drug treatment (> one week treatment);
* Laboratory values more than 15% outside the normal range for transaminases, CRP or bleeding parameters;
* Individuals with organic brain syndrome;
* Individuals who are taking anticoagulants;
* Individuals who are taking omega-3 supplements, currently or within 8 weeks of being included in the trial;
* Individuals who have other, severe, intercurrent illness which in the opinion of the investigator may put them at risk or influence the results of the trial.

Ages: 12 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure for this study is the transition to psychosis rate measured by the Comprehensive Assessment of At Risk Mental States (CAARMS) (Yung et al., 2005), | The time frame for the first outcome measure will be over the 12-month follow-up period.
  Transition to psychosis is operationally defined, based on the CAARMS (Yung et al., 2005) criteria: 1./Abnormal thoughts held with delusional intensity occurring every day for one week or longer; 2./True hallucinations in any modality occurring every day for one week or longer; or 3./Formal thought disorder to the degree of incoherence and/or loose associations occurring every day for one week or longer

SECONDARY OUTCOMES:
The secondary outcome measures are the transition to psychosis rate measured by the CAARMS, the Positive and Negative Syndrome Scale (PANSS), the Montgomery-Asberg Depression Rating Scale (MADRS) and the Global Assessment of Functioning Scale (GAF) | These scales will be performed at baseline, 4, 8, 12, 26, and 52 weeks.
  These instruments are widely used clinical scales for psychotic patients and guarantee standardized assessment when used with interview guides and operationalized anchor points.
Side effects of therapeutic interventions will be assessed using the UKU side effect rating scale (Lingjaerde et al., 1987). | Side effects will be assessed at baseline, 4, 8, 12, 26, and 52 weeks
Wechsler Adult Intelligence Scales-Revised, the Wechsler Memory Scale-Revised, the Wisconsin Card Sorting Test, Trail Making Test-Part A and B, the Continuous Performance Test, and the Finger Tapping Test: right and left | The neuropsychological battery will be performed at baseline and after 12 weeks (pre/post study design) and at 12 months follow-up.
  In accordance with Bilder et al. (2000) assessments will cover following neuropsychological functions: (1) memory (spatial short term memory, spatial working memory, visuospatial paired associate learning, pattern recognition, spatial recognition, delayed matching to sample), (2) executive, (3) attention, (4) language, (5) motor, (6) visuospatial.
Blood samples: EDTA blood in standard glass tubes (no plastic tubes because of artifacts for omega-3 PUFA analysis) | At baseline and after twelve weeks
  Blood samples will be collected and centrifuged as soon as possible at 1500g for 15 minutes. inPLA2 sample: 1 tube (5ml) EDTA blood: Plasma, buffy coat and the top 2 mm of RBCs will be aspirated and frozen. Omega-3 PUFA sample: 1 tube (10ml) EDTA blood: second wash step required. Samples will be frozen at -80 degrees Celsius.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Armando, MD, PhD, Principal Investigator — Bambino Gesù Hospital and Research Institute
Locations (1):
- Bambino Gesù Hospital and Research Institute, Vatican City, Vatican City State, Holy See